CLINICAL TRIAL: NCT02126046
Title: Unrelated Umbilical Cord Blood Following HLA-haploidentical Hematopoietic Stem Cell Transplantation in Patients With β-thalassemia Major
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Principal Investigator, Chunfu Li, Director and professor, Nanfang Hospital, Southern Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NFTM20130101
Record Dates: First submitted 2014-04-18; First posted 2014-04-29 (Estimated); Last update posted 2015-04-16 (Estimated); Status verified 2015-04

CONDITIONS: Thalassemia Major
Keywords: Cord Blood Transplant; Haploidentical HSCT; Thalassemia major
MeSH Terms: conditions — beta-Thalassemia

ARMS (1):
- Hi-HSC-CBT (Other)
  Interventions: Genetic: unrelated CB following haplo-identical hematopoietic stem cells transplantation

INTERVENTIONS:
Genetic: unrelated CB following haplo-identical hematopoietic stem cells transplantation

SUMMARY:
Allo-hematopoietic stem cell transplantation(HSCT) is the only way to cure β-thalassemia major at present. To expand donor pool，we developed a haplo-identical HSCT (Hi-HSCT) platform. But in prior Hi-HSCT using high dose post-transplant Cyclophosphamide in patients with leukemia, cytopenia post-transplant often developed, which was considered as a symptom of GVHD. Therefore, the investigators add unrelated umbilical cord blood (UCB) to the Hi-HSCT. It has reported that, as third-party cells, UCB will reduce GVHD.The purpose of this study is to determine whether unrelated UCB following Hi-HSCT can improve outcomes of Hi-HSCT in patients with β-thalassemia major.

ELIGIBILITY:
Inclusion Criteria:

* β-thalassemia major
* < 18 year old
* Unrelated umbilical cord blood following Haplo-identical HSCT

Exclusion Criteria:

* ≥ 18 year old
* HLA- matched related donors
* Unrelated donor transplants
* Unrelated umbilical cord blood transplants
* Severe iron overload in heart by T2*

Ages: 12 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2012-09; Primary Completion 2015-12 (Estimated); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
overall survival（OS） | 12 months
  the measure is a composite
TM-free survival（TFS） | 12 months
  the measure is a composite
Transplant Related Martality (TRM) | 12 months
  the measure is a composite
Primary or Secondary Graft Rejection (GR) | 12 months
  the measure is a composite

SECONDARY OUTCOMES:
The cumulative incidences of acute graft-versus-host disease（GVHD） | 12 months
  the measure is a composite
The cumulative incidences of chronic graft vesus host disease (cGVHD) | 12 months
  the measure is a composite

CONTACTS AND LOCATIONS:
Locations (1):
- Department of paediatrics，Nangfang Hospital, Southern Medical University, Guangzhou, Guangdong, China